CLINICAL TRIAL: NCT06738212
Title: Comparative Effects of Aerobic and Aviva Exercises on Pain Quality of Life, Sleep and Daily Functioning in Primary Dysmenorrhea
Brief Title: Comparative Effects of Aerobic and Aviva Exercises in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah international universit
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dysmenorrhea Primary
Keywords: Exercise; Quality of life; Sleep; Pain
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: A sample will be divided into two groups, each group will have 21 participants. The group A will be given Aerobic exercise and Group B will be given Aviva exercises.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercises (Experimental)
  Interventions: Other: Group A aerobic exercises
- Aviva Exercises (Active Comparator)
  Interventions: Other: Group B Aviva exercises

INTERVENTIONS:
Other: Group A aerobic exercises — Group A will perform the aerobic exercises (such as bicycling, treadmill and running) Aerobic exercises 15min/session for each exercise, 2 times/week. Frequency: 2 times /week Intensity: Easy to moderate about 60 to 75% of maximum heart rate Type: treadmill, bicycling, running Time: 45min/session
  Bicycling:
  15
  - Start with gentle, low-intensity cycling and gradually increase as comfort allows - Aim for regular, consistent cycling sessions (e.g., 2-3 times a week,15min/session) - Consider incorporating other exercises, like stretching or yoga, to complement cycling.
  Running
  To get started with running for dysmenorrhea:
  1. Start with short distances and gradually increase as comfort allows
  2. Aim for regular, consistent running sessions (e.g., 2-3 times a week,15 minute/session)
  3. Consider incorporating other exercises, like stretching or yoga, to complement running.
  Arms: Aerobic Exercises
Other: Group B Aviva exercises — Group B will perform the Aviva exercises in 18 different movements. Aviva exercise intervention method is based on a carefully structured, mild-to-moderate intensity series of 18 movement sequences and aerobic exercises 30min/session, 2 times/week (20)
  Aviva Methods of exercises:
  These exercises are a carefully structured, intense, and methodical series of movement sequences, including a 5 min warm-up exercise at the beginning and 5 min cooling-down exercises at the end of the session. These exercises are performed in Standing, Sitting, Supine lying, prone lying
  Arms: Aviva Exercises

SUMMARY:
Primary dysmenorrhea is a cramping pain in the lower abdomen occurring just before or during menstruation without pelvic pathology. Primary dysmenorrhea is not a life-threatening condition and does not cause organ failure. However, it can affect the quality of life of women and cause inability to carry out daily functioning consequently, absence from school or workplace. Exercise is one of the non-conservative methods to reduce the severity of primary dysmenorrhea. The aim of this study is to compare the effects of aerobic and Aviva exercises on primary dysmenorrhea. This study emphasizes the importance of aerobic exercises and Aviva exercise to reduce the severity of primary Dysmenorrhea. This will help in patients over all recovery and will improve general well-being.

This will be a Randomized clinical trial conducted on 42 participants. The data will be collected from Sharif Medical Complex and Kasrat Gym Lake City by using non-probability convenience sampling technique. Patients with primary dysmenorrhea diagnosed with Walid score questionnaire of age 20-40 will be included. A sample will be divided into two groups, each group will have 21 participants. The group A will be given Aerobic exercise and Group B will be given Aviva exercises. Participants will be assessed using the Mc Gill pain questionnaire for pain, women health initiative insomnia rating scale will be used for sleep, and brief pain inventory short form for daily functioning and Quality of life enjoyment and satisfaction questionnaire short form for quality of life. Data will be analyzed by using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried females
* Regular menstrual cycles (every 21-35 days)
* Moderate to severe menstrual cramp pain

Exclusion Criteria:

* Pelvic pathology (endometriosis, chronic pelvic inflammatory disease, adenomyosis)
* History of pelvic surgery or inflammatory disease
* Chronic pain or pain disorders (e.g., fibromyalgia)
* Current use of pain medication or muscle relaxants
* History of mental health disorders (e.g., depression, anxiety)
* Inability to understand or complete study assessments
* Any underlying medical condition that may be contributing to dysmenorrhea (e.g., thyroid disorders, kidney disease)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females suffering from PRIMARY DYSMENORRHEA
Enrollment: 42 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Mc Gill Pain Questionnaire | 12 weeks
  The Mc Gill pain questionnaire can be used to evaluate a person experiencing significant pain. It can be used to monitor the pain over time and to determine the effectiveness of any intervention.
  Validity and reliability 0.79 and 0.89.
Women's Health Initiative Insomnia Rating Scale (WHIIRS) | 12 weeks
  A brief five-item scale evaluating insomnia symptoms, the WHIIRS was developed as part of a larger study investigating a range of health issues affecting postmenopausal women. The scale requires individuals to rate the quality of their sleep and the frequency with which they experience certain sleep problems, providing a total score that may be useful for both research and clinical purposes.
Brief Pain Inventory Short Form SF 12 | 12 weeks
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is given the bidirectional link between sleep and pain. The range of the scale from 0 to 10.the internal reliability ranging from .95 to .97 for surgical cancer and .82 to .95 ranging for patient with low back pain and arthritis. It is often used as a quality-of-life measure.
Quality of Life Enjoyment and Satisfaction Questionnaire Short Form(Q-LES-Q-SF) | 12 weeks
  Quality of life Enjoyment and Satisfaction Questionnaire Short form evaluates general activities that are assessed in the longer form of the Q- LES-Q. Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good).

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Sharif Medical Complex & Kasrat gym, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anis T, Hasan S, Lohana N, Salahuddin I, Saeed HJJoXaSU, Natural Sciences Edition. Effects of aerobic program on the severity of dysmenorrhea using WaLIDD score. 2023;19(6):550-4
- [Background] Kovacs Z, Atombosiye E, Hegyi G, Szoke H. The Effect of Aviva Exercise Intervention on Pain Level and Body Awareness in Women with Primary Dysmenorrhea. Medicina (Kaunas). 2024 Jan 20;60(1):184. doi: 10.3390/medicina60010184. PMID 38276063
- [Background] Elbandrawy AM, Elhakk SM. Comparison between the effects of aerobic and isometric exercises on primary dysmenorrhea. 2021
- [Background] Gohil K, Mehta B. Effect of aerobic exercise on pain and quality of life in women with primary dysmenorrhea. International Journal of Applied Research. 2022;8(6):256-8
- [Background] Mohebbi Dehnavi Z, Jafarnejad F, Sadeghi Goghary S. The effect of 8 weeks aerobic exercise on severity of physical symptoms of premenstrual syndrome: a clinical trial study. BMC Womens Health. 2018 May 31;18(1):80. doi: 10.1186/s12905-018-0565-5. PMID 29855308